CLINICAL TRIAL: NCT01202032
Title: Bevacizumab in Patients With Metastatic Renal Cell Carcinoma or Others Advanced Solid Tumors
Brief Title: Multicenter Dose-escalation Study of a Combination of Pazopanib and Bevacizumab in Patients With Metastatic Renal Cell Carcinoma or Others Advanced Solid Tumors
Acronym: PARASOL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARASOL
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Renal Cell Carcinoma; Advanced Refractory Solid Tumors Histologically or Cytologically Confirmed
Keywords: Metastatic renal cell carcinoma; Advanced solid tumors; Dose escalation; Association Pazopanib-Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Association of Bevacizumab (BVC)+ Pazopanib (PZP) — Treatment is administered in 28-day cycles, during which patients received BVC intravenously every 2 weeks and oral PZP once daily from days 1 to 28. For the first cycle, PZP is administered alone from days 1 to 14.
  The starting dose for dose escalation is BVC at 7.5 mg/kg in combination with PZP 400 mg (level 1).
  The therapy regimens for each dose level are respectively:
  BVC 7.5 mg/kg + PZP 600 mg (level 2) BVC 10 mg/kg + PZP 600 mg (level 3) BVC 10 mg/kg + PZP 800 mg (level 4). Patients who experience grades 3 to 4 adverse events have dose adjustments to one or both drugs. Dose reductions affect in priority the administration of PZP. Doses reductions to PZP are made in 200-mg decrements and to BVC to 2.5-mg/kg decrements.
  Patients with toxicities that warrant reductions at either PZP 400 mg or BVC 7.5 mg/kg are withdrawn from the study.

SUMMARY:
This is an open-label, multicenter dose-escalation phase I study using a 3+3+3 design (i.e., 3 to 9 patients per dose level) in patients with mRCC or others advanced refractory solid tumors. Enrolment will be performed to include approximately ½ of patients with mRCC.

The primary endpoint is the occurrence of limiting toxicities leading to definitive discontinuation of the study drugs during the first 24 weeks in absence of progression of the disease.

Secondary endpoints included the occurrence of Dose Limiting Toxicities (DLTs) evaluated during the first two cycles; overall response rate, 6-months progression-free survival rate and Pharmacokinetic assessments.

DETAILED DESCRIPTION:
The primary endpoint is the occurrence of limiting toxicities leading to definitive discontinuation of the study drugs during the first 24 weeks in absence of progression of the disease.

Secondary endpoints included the occurrence of Dose Limiting Toxicities (DLTs) evaluated during the first two cycles; overall response rate (ORR), 6-months progression-free survival rate and Pharmacokinetic assessments.

The following definitions will be used:

DLT:

The Dose Limiting Toxicities (DLTs) are defined as the occurrence during the first two cycles of any grade 4 toxicity, and of any following events:

* clinical evidence of congestive heart failure,
* any arterial thromboembolic event,
* grade 3 venous thrombosis,
* grade 3 thrombocytopenia >=7 days or associated with bleeding,
* grade 3 hypertension uncontrolled (>=160/90 mmHg) with medications,
* grade 3 elevations in AST/ALT or total bilirubin. Any other grade 3 toxicity >=7 days is also considered as a DLT, with exception of fatigue.

MTD:

The determination of the maximum-tolerated dose (MTD) will be conducted on a 3 + 3 + 3 design. Cohorts of 3 to 9 patients will be sequentially enrolled in 3 steps to receive one of four escalated doses of Pazopanib in combination with Bevacizumab to establish the MTD (step 1: patients 1 to 3; step 2: patients 4 to 6; step 3: patients 7 to 9).

The MTD is considered to be exceeded if DLT is observed during the first 2 cycles (i.e., 56 days) in at least 2 out of 3 or 3 out of 6 patients evaluable for MTD in the two first steps, then in at least 3 out of 9 patients after completion of enrolment (step 3).

When the MTD will be established, patients already involved in the follow-up phase at a dose level above the MTD should decrease to the MTD.

Note: in an exploratory way (i.e., with simulation) the possibility to take into account for the determination of the MTD the occurrence of recurrent grade 2 events or the combination of synergic grade 2-3 toxicities as "1/2 DLT" will be investigated in the study.

Optimal Long Exposure Dose (OLED):

To determine the Optimal Long Exposure Dose (OLED), all patients which will not experience a Dose Limiting Toxicity (DLT) during the first two cycles will continue the treatment and will be followed until week 24, in order to record toxic reactions of lesser severity or mixed toxicities leading to definitive discontinuation of the study drug, in the absence of progression of the disease.

The OLED is defined as the dose level (less than or equal to the MTD) for which the occurrence of sub-acute limiting toxicities leading to definitive discontinuation of the study drug is compatible with further phase II studies.

In practice, if <=2/7-8 patients or <=3/9 patients treated at a dose level <=MTD and followed until week 24 experience sub-acute limiting toxicities, that dose level will be considered as the OLED.

ORR:

The overall response rate (ORR) is defined as the proportion of patients with a complete response (CR) or partial response (PR) - target lesions and tumor response according to RECIST guidelines.

Progression-Free Survival (PFS):

Progression-free survival (PFS) is defined as the time from the date of first study drug administration to the date of the first observation of documented disease progression or death due to any cause. PFS will be determined based on tumor assessment (RECIST criteria) and survival information.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Dated and signed written informed consent.
* Histologically progressive mRCC or other advanced refractory histologically or cytologically confirmed solid tumors. In mRCC situation, only patients who have received no prior therapy or who have failed only one prior systemic therapy (except tyrosine kinase inhibitors) are allowed; for patients with other advanced refractory solid tumors, no more than three prior systemic therapy regimens (except tyrosine kinase inhibitors) are permitted.
* ECOG performance status of 0 or 1.
* At least one measurable site of disease as defined by RECIST criteria 1.1. based on investigator's assessment.
* Adequate bone marrow function: absolute neutrophil count >=1.5 x 109/L, platelet count >= 100 x 109/L, and hemoglobin >= 9 g/dL.
* Adequate liver function: AST/ALT <= 2 x upper limit of normal (ULN) and total bilirubin in the normal values.
* Adequate coagulation function: prothrombin time (PT) or international normalized ratio (INR) <=1.2 x ULN and activated partial thromboplastin time (APTT)<=1.2x ULN.
* Adequate renal function: serum creatinine ≤ 1.5 mg/dL (133 µmol/L) or, if greater than 1.5 mg/dL: calculated creatinine clearance ≥ 50 mL/min.
* Absence of proteinuria confirmed by urinary dipstick test. If the dipstick test is twice positive, proteinuria will be quantified on a complete 24h urine sample: urine protein value must be <1 g /L.
* Ability to swallow and retain oral medication.
* Adequate contraception methods.
* Mandatory affiliation with a health insurance company.

Exclusion Criteria:

* Prior Pazopanib treatment.
* Prior Bevacizumab treatment within 6 months prior to begin study treatment. Patients with any grade 3 or grade 4 toxicity during prior BVC therapy are not eligible.
* Prior treatment with any tyrosine kinase inhibitor.
* Concomitant participation to an other clinical study estimating a experimental agent.
* Patients with any haematological, renal, or neurological grade 3-4 toxicity during prior systemic therapy regimens.
* Patients with any liver injury grade 3-4 during prior systemic therapy regimens.
* Patients with squamous non-small cell lung carcinoma.
* Patients with high vascular and nephrologic risks [uncontrolled hypertension while receiving appropriate medication (SBP ≥ 150 mmHg and DBP ≥ 90 mmHg), significant proteinuria, low creatinine clearance level…].
* Patients with brain metastases.
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing:

Active peptic ulcer disease;kown intraluminal metastatic lesion/s with suspected bleeding;inflammatory bowel disease; ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment; malabsorption syndrome; major resection of the stomach or small bowel.

* History of Gilbert's disease.
* Patients with chronic hepatitis.
* Any unstable or serious concurrent condition (i.e., presence of uncontrolled infection).
* Prolongation of corrected QT interval (QTc) >480 msecs using Bazett's formula.
* History of any one of more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting; myocardial infarction; unstable angina; symptomatic peripheral vascular disease; coronary artery by-pass graft surgery; class III or IV congestive heart failure as defined by the New York Heart Association (NYHA); history of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulant agents (excluding therapeutic warfarin) for at least 6 weeks are eligible.

* Hemoptysis within 6 weeks of first dose of study drug.
* Evidence of active bleeding or bleeding diathesis.
* Anticoagulant treatment with curative intent.
* Known endobronchial lesions or involvement of large pulmonary vessels by tumor.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Radiation therapy, surgery or tumor embolization within 2 weeks prior to the first dose of study drug.
* Chemotherapy, immunotherapy, biological therapy, hormonal therapy or treatment with an investigational agent within 14 days or 5 half-lives, whichever is longer prior to the first dose of study drug.
* Patient unable or unwilling to discontinue predefined prohibited medications listed in the protocol for 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to PZP.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Clinically assessed as having inadequate venous access for PK sampling.
* Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determination of the Optimal Long Exposure Dose (OLED) | 24 weeks for each patient
  The primary endpoint is the occurrence of an interruption of one drug of the association of a duration superior to 4 weeks during the first 24 weeks in absence of progression of the disease.

SECONDARY OUTCOMES:
The determination of the maximum-tolerated dose (MTD) | 8 weeks for each patient
To estimate the overall response rate (ORR) | 24 weeks
To estimate the 6-month progression-free survival (PFS) rate | 24 weeks
To characterize the pharmacokinetic (PK) profile of Pazopanib when combined with Bevacizumab. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SYLVIE NEGRIER, Phd, Principal Investigator — Centre Léon Bérard; Lyon; FRANCE
Locations (1):
- Centre Léon BERARD, Lyon, France

REFERENCES:
- [Background] Ferrara N, Gerber HP, LeCouter J. The biology of VEGF and its receptors. Nat Med. 2003 Jun;9(6):669-76. doi: 10.1038/nm0603-669. PMID 12778165
- [Background] Dvorak HF. Vascular permeability factor/vascular endothelial growth factor: a critical cytokine in tumor angiogenesis and a potential target for diagnosis and therapy. J Clin Oncol. 2002 Nov 1;20(21):4368-80. doi: 10.1200/JCO.2002.10.088. PMID 12409337
- [Background] Kumar R, Knick VB, Rudolph SK, Johnson JH, Crosby RM, Crouthamel MC, Hopper TM, Miller CG, Harrington LE, Onori JA, Mullin RJ, Gilmer TM, Truesdale AT, Epperly AH, Boloor A, Stafford JA, Luttrell DK, Cheung M. Pharmacokinetic-pharmacodynamic correlation from mouse to human with pazopanib, a multikinase angiogenesis inhibitor with potent antitumor and antiangiogenic activity. Mol Cancer Ther. 2007 Jul;6(7):2012-21. doi: 10.1158/1535-7163.MCT-07-0193. PMID 17620431
- [Background] Hutson TE, Davis ID, Machiels JP, De Souza PL, Rottey S, Hong BF, Epstein RJ, Baker KL, McCann L, Crofts T, Pandite L, Figlin RA. Efficacy and safety of pazopanib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2010 Jan 20;28(3):475-80. doi: 10.1200/JCO.2008.21.6994. Epub 2009 Dec 14. PMID 20008644
- [Background] Escudier B, Pluzanska A, Koralewski P, Ravaud A, Bracarda S, Szczylik C, Chevreau C, Filipek M, Melichar B, Bajetta E, Gorbunova V, Bay JO, Bodrogi I, Jagiello-Gruszfeld A, Moore N; AVOREN Trial investigators. Bevacizumab plus interferon alfa-2a for treatment of metastatic renal cell carcinoma: a randomised, double-blind phase III trial. Lancet. 2007 Dec 22;370(9605):2103-11. doi: 10.1016/S0140-6736(07)61904-7. PMID 18156031
- [Background] Rini BI, Halabi S, Rosenberg JE, Stadler WM, Vaena DA, Ou SS, Archer L, Atkins JN, Picus J, Czaykowski P, Dutcher J, Small EJ. Bevacizumab plus interferon alfa compared with interferon alfa monotherapy in patients with metastatic renal cell carcinoma: CALGB 90206. J Clin Oncol. 2008 Nov 20;26(33):5422-8. doi: 10.1200/JCO.2008.16.9847. Epub 2008 Oct 20. PMID 18936475
- [Background] Belot A, Grosclaude P, Bossard N, Jougla E, Benhamou E, Delafosse P, Guizard AV, Molinie F, Danzon A, Bara S, Bouvier AM, Tretarre B, Binder-Foucard F, Colonna M, Daubisse L, Hedelin G, Launoy G, Le Stang N, Maynadie M, Monnereau A, Troussard X, Faivre J, Collignon A, Janoray I, Arveux P, Buemi A, Raverdy N, Schvartz C, Bovet M, Cherie-Challine L, Esteve J, Remontet L, Velten M. Cancer incidence and mortality in France over the period 1980-2005. Rev Epidemiol Sante Publique. 2008 Jun;56(3):159-175. doi: 10.1016/j.respe.2008.03.117. Epub 2008 Jun 10. PMID 18547762
- [Background] Remontet L, Esteve J, Bouvier AM, Grosclaude P, Launoy G, Menegoz F, Exbrayat C, Tretare B, Carli PM, Guizard AV, Troussard X, Bercelli P, Colonna M, Halna JM, Hedelin G, Mace-Lesec'h J, Peng J, Buemi A, Velten M, Jougla E, Arveux P, Le Bodic L, Michel E, Sauvage M, Schvartz C, Faivre J. Cancer incidence and mortality in France over the period 1978-2000. Rev Epidemiol Sante Publique. 2003 Feb;51(1 Pt 1):3-30. PMID 12684578
- [Background] Diaz JI, Mora LB, Hakam A. The Mainz Classification of Renal Cell Tumors. Cancer Control. 1999 Nov;6(6):571-579. doi: 10.1177/107327489900600603. PMID 10756388
- [Background] Nelson EC, Evans CP, Lara PN Jr. Renal cell carcinoma: current status and emerging therapies. Cancer Treat Rev. 2007 May;33(3):299-313. doi: 10.1016/j.ctrv.2006.12.005. Epub 2007 Feb 27. PMID 17329029
- [Background] Lam JS, Belldegrun AS, Pantuck AJ. Long-term outcomes of the surgical management of renal cell carcinoma. World J Urol. 2006 Aug;24(3):255-66. doi: 10.1007/s00345-006-0055-5. Epub 2006 Feb 15. PMID 16479388
- [Background] Mickisch G, Carballido J, Hellsten S, Schulze H, Mensink H; European Association of Urology. Guidelines on renal cell cancer. Eur Urol. 2001 Sep;40(3):252-5. doi: 10.1159/000049783. PMID 11684839
- [Background] Yagoda A, Abi-Rached B, Petrylak D. Chemotherapy for advanced renal-cell carcinoma: 1983-1993. Semin Oncol. 1995 Feb;22(1):42-60. No abstract available. PMID 7855619
- [Background] Negrier S, Perol D, Ravaud A, Chevreau C, Bay JO, Delva R, Sevin E, Caty A, Escudier B; French Immunotherapy Intergroup. Medroxyprogesterone, interferon alfa-2a, interleukin 2, or combination of both cytokines in patients with metastatic renal carcinoma of intermediate prognosis: results of a randomized controlled trial. Cancer. 2007 Dec 1;110(11):2468-77. doi: 10.1002/cncr.23056. PMID 17932908
- [Background] Negrier S, Perol D, Ravaud A, Bay JO, Oudard S, Chabaud S, Fargeot P, Delva R, Deplanque G, Gravis G, Escudier B; French Immunotherapy Group. Randomized study of intravenous versus subcutaneous interleukin-2, and IFNalpha in patients with good prognosis metastatic renal cancer. Clin Cancer Res. 2008 Sep 15;14(18):5907-12. doi: 10.1158/1078-0432.CCR-08-0236. PMID 18794104
- [Background] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Oudard S, Negrier S, Szczylik C, Pili R, Bjarnason GA, Garcia-del-Muro X, Sosman JA, Solska E, Wilding G, Thompson JA, Kim ST, Chen I, Huang X, Figlin RA. Overall survival and updated results for sunitinib compared with interferon alfa in patients with metastatic renal cell carcinoma. J Clin Oncol. 2009 Aug 1;27(22):3584-90. doi: 10.1200/JCO.2008.20.1293. Epub 2009 Jun 1. PMID 19487381
- [Background] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- [Background] Ellis LM, Hicklin DJ. VEGF-targeted therapy: mechanisms of anti-tumour activity. Nat Rev Cancer. 2008 Aug;8(8):579-91. doi: 10.1038/nrc2403. Epub 2008 Jul 3. PMID 18596824
- [Background] Azad NS, Posadas EM, Kwitkowski VE, Steinberg SM, Jain L, Annunziata CM, Minasian L, Sarosy G, Kotz HL, Premkumar A, Cao L, McNally D, Chow C, Chen HX, Wright JJ, Figg WD, Kohn EC. Combination targeted therapy with sorafenib and bevacizumab results in enhanced toxicity and antitumor activity. J Clin Oncol. 2008 Aug 1;26(22):3709-14. doi: 10.1200/JCO.2007.10.8332. PMID 18669456
- [Background] Rini BI, Garcia JA, Cooney MM, Elson P, Tyler A, Beatty K, Bokar J, Mekhail T, Bukowski RM, Budd GT, Triozzi P, Borden E, Ivy P, Chen HX, Dolwati A, Dreicer R. A phase I study of sunitinib plus bevacizumab in advanced solid tumors. Clin Cancer Res. 2009 Oct 1;15(19):6277-83. doi: 10.1158/1078-0432.CCR-09-0717. Epub 2009 Sep 22. PMID 19773375
- [Background] Feldman DR, Baum MS, Ginsberg MS, Hassoun H, Flombaum CD, Velasco S, Fischer P, Ronnen E, Ishill N, Patil S, Motzer RJ. Phase I trial of bevacizumab plus escalated doses of sunitinib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2009 Mar 20;27(9):1432-9. doi: 10.1200/JCO.2008.19.0108. Epub 2009 Feb 17. PMID 19224847
- [Background] Katavetin P, Katavetin P. VEGF inhibition and renal thrombotic microangiopathy. N Engl J Med. 2008 Jul 10;359(2):205-6; author reply 206-7. doi: 10.1056/NEJMc080770. No abstract available. PMID 18614790
- [Background] Ratain MJ, Sargent DJ. Optimising the design of phase II oncology trials: the importance of randomisation. Eur J Cancer. 2009 Jan;45(2):275-80. doi: 10.1016/j.ejca.2008.10.029. Epub 2008 Dec 6. PMID 19059773
- [Background] Motzer RJ, Bacik J, Murphy BA, Russo P, Mazumdar M. Interferon-alfa as a comparative treatment for clinical trials of new therapies against advanced renal cell carcinoma. J Clin Oncol. 2002 Jan 1;20(1):289-96. doi: 10.1200/JCO.2002.20.1.289. PMID 11773181
- [Background] Coppin C, Porzsolt F, Awa A, Kumpf J, Coldman A, Wilt T. Immunotherapy for advanced renal cell cancer. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001425. doi: 10.1002/14651858.CD001425.pub2. PMID 15674877
- [Background] Coppin C, Le L, Porzsolt F, Wilt T. Targeted therapy for advanced renal cell carcinoma. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD006017. doi: 10.1002/14651858.CD006017.pub2. PMID 18425931
- [Derived] Negrier S, Perol D, Bahleda R, Hollebecque A, Chatelut E, Boyle H, Cassier P, Metzger S, Blanc E, Soria JC, Escudier B. Phase I dose-escalation study of pazopanib combined with bevacizumab in patients with metastatic renal cell carcinoma or other advanced tumors. BMC Cancer. 2017 Aug 15;17(1):547. doi: 10.1186/s12885-017-3527-7. PMID 28810837
- [Derived] Imbs DC, Negrier S, Cassier P, Hollebecque A, Varga A, Blanc E, Lafont T, Escudier B, Soria JC, Perol D, Chatelut E. Pharmacokinetics of pazopanib administered in combination with bevacizumab. Cancer Chemother Pharmacol. 2014 Jun;73(6):1189-96. doi: 10.1007/s00280-014-2455-3. Epub 2014 Apr 6. PMID 24705975
- See also: Related Info — http://seer.cancer.gov/csr/1975_2005/